CLINICAL TRIAL: NCT02697149
Title: The Effectiveness and Safety of Nonradiation-to-endoscopist Endoscopic Retrograde Cholangiopancreatography in Patients With Complexity Level I/II
Brief Title: Nonradiation-to-endoscopist Endoscopic Retrograde Cholangiopancreatography in Patients With Complexity Level I/II
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: 20151203-5
Record Dates: First submitted 2015-12-17; First posted 2016-03-03 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography , Gallstone
Keywords: ERCP; nonradiation-to-endoscopist; gallstones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- intervention: patients undergoing nonradiation-to-endoscopist endoscopic retrograde cholangiopancreatography
  Interventions: Radiation: nonradiation-to-endoscopist endoscopic retrograde cholangiopancreatography
- control: patients undergoing standard endoscopic retrograde cholangiopancreatography
  Interventions: Radiation: standard endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Radiation: nonradiation-to-endoscopist endoscopic retrograde cholangiopancreatography — All patients received magnetic resonance cholangiopancreatography before the procedure. Characteristics of lesions (e.g. common bile duct stones, stenosis) in detail was identified. During the procedure, the endoscopist was not exposed to radiation. If fluoroscopy was needed, after contrast injection (sometimes not necessary), the endoscopist went outside of the operation room and observed the X-ray image by remote control of the fluoroscopy machine.
  Groups: intervention
Radiation: standard endoscopic retrograde cholangiopancreatography — Patients received standard endoscopic retrograde cholangiopancreatography. Fluoroscopy was normally used when necessary.
  Groups: control

SUMMARY:
Radiation exposure may put endoscopists at risk when performing endoscopic retrograde cholangiopancreatography. Although non-radiation endoscopic retrograde cholangiopancreatography was reported in pregnant women in previous reports, it remains unclear whether endoscopic retrograde cholangiopancreatography is also effective and safe when endoscopists were not expose to radiation. This study was to evaluate the effectiveness and safety of nonradiation-to-endoscopist endoscopic retrograde cholangiopancreatography in patients with complexity level I/II.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old
* patients undergoing endoscopic retrograde cholangiopancreatography

Exclusion Criteria:

* 1 Bismuth typy Ⅲ and Ⅳ
* 2 common bile duct stone > 15mm
* 3 common bile duct stone and distal stenosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-90 years old, patients undergoing endoscopic retrograde cholangiopancreatography
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Success of endoscopic retrograde cholangiopancreatography | 6 months
  The success is defined by complete removal of common bile duct stones or placement of stents in proper position.

SECONDARY OUTCOMES:
Overall complications | 6 months
  Post-endoscopic retrograde cholangiopancreatography pancreatitis, bleeding, perforation, infection of biliary tract
Cannulation success rate | 6 months
  In patients with native papilla, cannulation success rate was defined as the proportion of subjects with successful cannulation of targeted duct
ERCP procedure time | 6 months
  defined by the interval time between scope insertion and complete of endoscopic retrograde cholangiopancreatography

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Air Force Military Medical University, China; Wei Zeng, M.D., Principal Investigator — Department of gastroenterology, Chinese PLA 174 hospital
Locations (2):
- China (2):
  - Department of gastroenterology, Chinese PLA 174 Hospital, Xiamen, Fujian
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Background] Uradomo LT, Goldberg EM, Darwin PE. Time-limited fluoroscopy to reduce radiation exposure during ERCP: a prospective randomized trial. Gastrointest Endosc. 2007 Jul;66(1):84-9. doi: 10.1016/j.gie.2006.10.055. PMID 17591479
- [Result] Liao C, Thosani N, Kothari S, Friedland S, Chen A, Banerjee S. Radiation exposure to patients during ERCP is significantly higher with low-volume endoscopists. Gastrointest Endosc. 2015 Feb;81(2):391-8.e1. doi: 10.1016/j.gie.2014.08.001. Epub 2014 Oct 5. PMID 25293825